CLINICAL TRIAL: NCT05176574
Title: Identification of Knowledge, Attitudes, Intensions, Abilities and Behavior on Physicians Who Manage Patients With Chronic, Non-communicable Diseases on Physical Activity and Exercise.
Brief Title: Physicians' Perceptions on Physical Activity and Exercise in Non Communicable Diseases.
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Syrou Niki, RN,MPH, PhD, Laboratory Teaching Staff, University of Thessaly
Other Study IDs: NCDs-Physicians' Perceptions
Record Dates: First submitted 2021-11-19; First posted 2022-01-04 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Physicians' Perceptions on Physical Activity and Exercise for Health
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physicians: Physicians from 12 different specialties (i.e. General Medicine, Endocrinologists, Neurologists, Cardiologists, Orthopedists, Pathologists, Rheumatologists, Phytochemists-Pneumonologists, Vascular Surgeons, Oncologists-Pathologists, Psychiatrists, Neurologists-Psychiatrists) who manage patients with non-communicable diseases.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — A questionnaire will be developed via the Delphi method, will be pilot tested and implemented to assess physicians' perceptions and behaviors on physical activity and exercise in chronic, non-communicable diseases.

SUMMARY:
This descriptive, cross sectional study aims to investigate the knowledge, attitudes, intentions, abilities, and behavior of physicians who manage patients with chronic, non-communicable, diseases about physical activity and exercise. The sample will be nationwide and consisted of about 20.350 physicians of all the 13 Greek Regions. An anonymous, coded and self- administered questionnaire will be used as the main research tool for measuring the knowledge, attitudes, intentions, abilities and behavior of physicians. The questionnaire will be developed via the Delphi method after a systematic literature review and a focus group. The construction of the main questionnaire via the Delphi method, will include 2-3 quantitative rounds of data collection by 16 experts. The experts, who will be physicians and have knowledge and experience in matters related to physical activity, exercise and chronic diseases, will be selected based on specific criteria. Once the questionnaire has been developed, it will be piloted on a sample of approximately 40-50 physicians - different from that of the study. Then it will be sent to the physicians of the main study. Beside the main questionnaire, the Greek Edition of International Physical Activity Assessment Questionnaire (International Physical Activity Questionnaire-Short, IPAQ), will be also provided to the physicians to evaluate their levels of physical activity. Both the questionnaires will be completed online, via electronic form (google), because of the Covid-19 pandemic. The questionnaires and the information letter will be sent electronically to the participants through the Panhellenic Medical Association. This study has been approved by the Bioethics and Ethics Committee of the School of Medicine of National and Kapodistrian University of Athens.

DETAILED DESCRIPTION:
This nationwide, cross-sectional study aims at investigating the knowledge, attitudes, intentions, abilities and behavior of physicians who manage patients with chronic, non-communicable diseases on physical activity and exercise. Secondly, it aims at developing a new questionnaire via the Delphi method that evaluates the knowledge, attitudes, intentions, abilities, and behavior on physical activity and exercise of physicians who manage patients with non-communicable diseases, and be weighted in terms of its validity and reliability.

The study will be conducted in Greece, in three main phases: 1) development of a new research tool (questionnaire) based on the questions of a draft questionnaire generated from the results of a systematic literature review and a focus group between researchers. The new questionnaire will explore the knowledge, attitudes, intentions, abilities, and behavior of physicians who manage patients with non-communicable diseases on physical activity and exercise, 2) pilot testing of the new questionnaire, and 2) main study implementation.

Phase 1: Construction of the questionnaire via the Delphi method.

The purpose of the Delphi method is to reach a consensus / agreement on questions about physicians' knowledge, attitudes, intentions, abilities, and behavior regarding physical activity and exercise and the research question of the method is: "What are the questions with consensus≥75% that will be included in the final main study questionnaire, which will explore physicians' knowledge, attitudes, intentions, abilities, and behavior in physical activity and exercise? ".

Delphi method research design: A two or three-round Delphi survey, with a list of questions on physicians' knowledge, attitudes, intentions, abilities, and behavior (draft questionnaire) generated from the results of a systematic literature review and a focus group between researchers, will be conduct. The draft questionnaire will be provided by principal researcher to the Delphi experts in the 1st round of the method, as described below. Specifically, at the first round of the procedure the experts will be invited to participate to Delphi method via e-mail. The method will start after obtaining their informed consent. Then the principal researcher will send to experts, via a google form, an anonymous, self- administered, coded and semi-structured questionnaire (draft), with closed and open questions, on which experts must give their consensus. The definition for consensus is percent agreement, with 75% being the threshold to define consensus. There will be two defined criteria to terminate the Delphi method; the one is the achievement of consensus≥75% and the second is the specific number of rounds (maximum 3). The experts will score on a 7/Likert scale (from 1, completely insignificant question to 7, completely important question). Under each closed question there will be the same open optional question (comment/justify) for adding comments. As well, at the end of each section there will be an additional open-ended question, to suggest, if desired, their own questions for the next round questionnaire. The questions of the semi-structured questionnaire will be divided into 6 main sections: Demographic and educational characteristics, knowledge, attitudes, intentions, abilities and behavior in physical activity and exercise.

After the collection of the 1st round data, a statistical analysis of the answers will be conducted and the experts will be informed about the first results, in the context of their feedback. This will give them the opportunity to change their point of view if they wish. Based on the results of the 1st round, the research team will construct the semi-structured questionnaire of the 2nd round, which will be checked of its face validity. The 2nd round will be conducted 2-3 weeks after and in accordance with the 1st round. The data collection of the 2nd round will be followed by their statistical analysis, feedback and the creation of the final questionnaire, if the desired consensus will be reached. If it will not, then the questionnaire will be sent back to the experts in a 3rd and final round 2-3 weeks after the 2nd round. The implementation of the Delphi method is scheduled for 01/2022 to 03/2022.

Phase 2: Pilot implementation and weighting of the main new research tool (questionnaire).

After the Delphi method, the final questionnaire will be pilot tested on a sample of 40-50 physicians from the 12 specialties of the main study. The pilot test will be conducted to evaluate feasibility, duration, adverse events, and improve upon the study design prior to performance of the full-scale research. The implementation of the pilot study is scheduled for 04/2022 to 06/2022.

Phase 3: Implementation of the main study.

The main study aims to investigate the knowledge, attitudes, intentions, abilities and behavior regarding physical activity and exercise of physicians who manage patients with chronic, non-communicable, diseases. The sample will be nationwide and consisted of about 20.350 physicians of all the 13 Greek Regions. An anonymous, coded and self- administered questionnaire will be used as the main research tool for investigating the knowledge, attitudes, intentions, abilities and behavior of physicians. The questionnaire will be developed via the Delphi method after a systematic literature review and a focus group and will be pilot tested, according to the above mentioned. After its pilot testing, the questionnaire will be provided to the physicians of the main study for completion. Beside the main questionnaire, the Greek Edition of International Physical Activity Assessment Questionnaire (International Physical Activity Questionnaire-Short, IPAQ, 8 items), will be also provided to the physicians to evaluate their levels of physical activity. Both questionnaires will be completed online, via electronic form (google), because of the Covid-19 pandemic. The questionnaires and the information letter will be sent electronically (via email) to the participants through the Panhellenic Medical Association or the local Medical Associations. This study has been approved by the Bioethics and Ethics Committee of the School of Medicine of National and Kapodistrian University of Athens. The implementation of the main study is scheduled for 06/2022 to 02/2023.

ELIGIBILITY:
Inclusion Criteria:

* Physicians with specific specialties: General Medicine, Endocrinologists, Neurologists, Cardiologists, Orthopedists, Pathologists, Rheumatologists, Phytochemists-Pneumonologists, Vascular Surgeons, Oncologists-Pathologists, Psychiatrists, Neurologists-Psychiatrists.
* Physicians who are active members of the Panhellenic Medical Association.

Exclusion Criteria:

* Physicians with other specialties than those described above.
* Physicians who are not members of the Panhellenic Medical Association.

Ages: 28 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Greek physicians who are members of the Panhellenic Medical Association, have one of the following specialties: General Medicine, Endocrinologists, Neurologists, Cardiologists, Orthopedists, Pathologists, Rheumatologists, Phytochemists-Pneumonologists, Vascular Surgeons, Oncologists-Pathologists, Psychiatrists, Neurologists-Psychiatrists, and manage patients with chronic non-communicable diseases.
Sampling Method: Non-Probability Sample
Enrollment: 546 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Investigation of physicians' knowledge on physical activity and exercise via questionnaire. | Once during the third phase of the main study (i.e. from 06/2022 to 02/2023)
  Physicians' knowledge on physical activity and exercise will be assessed via questionnaire.
  Only physicians who manage patients with chronic, non-communicable diseases will be included.
Investigation of physicians' attitudes on physical activity and exercise via questionnaire | Once during the third phase of the main study (i.e. from 06/2022 to 02/2023)
  Physicians' attitudes on physical activity and exercise will be assessed via questionnaire.
  Only physicians who manage patients with chronic, non-communicable diseases will be included.
Investigation of physicians' intensions on physical activity and exercise via questionnaire | Once during the third phase of the main study (i.e. from 06/2022 to 02/2023)
  Physicians' intensions on physical activity and exercise will be assessed via questionnaire.
  Only physicians who manage patients with chronic, non-communicable diseases will be included.
Investigation of physicians' abilities on physical activity and exercise via questionnaire | Once during the third phase of the main study (i.e. from 06/2022 to 02/2023)
  Physicians' abilities on physical activity and exercise will be assessed via questionnaire.
  Only physicians who manage patients with chronic, non-communicable diseases will be included.
Investigation of physicians' behaviors on physical activity and exercise via questionnaire | Once during the third phase of the main study (i.e. from 06/2022 to 02/2023)
  Physicians' behaviors on physical activity and exercise will be assessed via questionnaire.
  Only physicians who manage patients with chronic, non-communicable diseases will be included.

SECONDARY OUTCOMES:
Investigation of physicians' demographic characteristics via questionnaire | Once during the third phase of the main study (i.e. from 06/2022 to 02/2023)
  Physicians' gender, age, family status, educational level, health status, occupational status, residence status will be assessed via questionnaire. Only physicians who manage patients with chronic, non-communicable diseases will be included.
Investigation of physicians' physical activity level | Once during the third phase of the main study (i.e. from 06/2022 to 02/2023)
  Physicians' weekly physical activity level will be assessed using the IPAQ questionnaire (short version). Only physicians who manage patients with chronic, non-communicable diseases will be included.

CONTACTS AND LOCATIONS:
Overall Officials: Niki Syrou, PhD, Principal Investigator — Department of Physical Education and Sport Science, University of Thessaly
Locations (1):
- Department of Physical Education and Sports Science, University of Thessaly, Trikala, Greece